CLINICAL TRIAL: NCT04013971
Title: Innovative Biofeedback Interface for Enhancing Stroke Gait Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Trisha Kesar, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00106866; 1R21HD095138-01 (NIH)
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Gait, Hemiplegic; Stroke
Keywords: stroke; gait rehabilitation; game
MeSH Terms: conditions — Gait Disorders, Neurologic; Stroke

STUDY DESIGN:
Intervention Model Description: This study aims to enroll 12 post-stroke and 12 able-bodied individuals who will complete gait trials with 2 different biofeedback interfaces in each experimental session.
Who Masked: Outcomes Assessor
Masking Description: The study outcomes will comprise objective biomechanical measures derived using motion capture, which will be processed by lab personnel who are blinded to the gait training condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-stroke Participants (Other): Post-stroke participants completing gait training trials with two different biofeedback interfaces in each experimental session. Participants also complete a control condition where no biofeedback is provided.
  Interventions: Other: AGRF Biofeedback Game; Other: Traditional Biofeedback Interface; Other: Control Condition
- Able-bodied Participants (Other): Able-bodied individuals completing gait training trials with two different biofeedback interfaces in each experimental session. Participants also complete a control condition where no biofeedback is provided.
  Interventions: Other: AGRF Biofeedback Game; Other: Traditional Biofeedback Interface; Other: Control Condition

INTERVENTIONS:
Other: AGRF Biofeedback Game — During the AGRF biofeedback game participants will walk on a split-belt treadmill with a projector or screen display. Participants will be receiving real-time information or feedback about ongoing gait performance parameters while they are walking. The participants will be exposed to the AGRF biofeedback game for 4 minutes.
  Other Names: gait training bout
Other: Traditional Biofeedback Interface — For the traditional non-game biofeedback, the visual display comprises a horizontal line graph with a moveable cursor that represents the current measured value of antero-posterior ground reaction force for the targeted leg. The auditory feedback comprises an audible "beep" produced every time the cursor entered the target range. Participants will be exposed to the traditional biofeedback interface for 4 minutes.
  Other Names: gait training
Other: Control Condition — Participants will complete a control walk with out feedback.

SUMMARY:
This study will conduct a preliminary evaluation of and obtain user data on a novel game-based visual interface for stroke gait training. Study participants will complete one session comprising exposure to gait biofeedback systems in an order determined by randomization. Participants will be exposed to 2 types of biofeedback interfaces:

* newly developed game-based interface (projector screen display)
* traditional, non-game interface

DETAILED DESCRIPTION:
Stroke is the leading cause of adult disability. Even after discharge from rehabilitation, residual gait deficits are prevalent in stroke survivors, leading to decreased walking speed and endurance. Because gait dysfunctions limit community mobility, stroke survivors and rehabilitation clinicians consider restoration of walking a major goal of rehabilitation. Several challenges and research gaps limit the effectiveness of current clinical gait rehabilitation practices. While there is consensus that stroke survivors benefit from gait rehabilitation, agreement is lacking on which specific training interventions are most efficacious. The long-term goal of this proposal is to address these challenges by developing personalized, engaging, salient gait training treatments founded on evidence from neuroscience, biomechanics, motor learning, and gaming.

Real-time biofeedback is a promising gait training intervention for targeting specific biomechanical impairments. Biofeedback can enhance an individual's awareness of the impairment targeted during gait training, enabling self-correction of aberrant gait patterns.

In response to treadmill training combined with visual and auditory real-time biofeedback, able-bodied individuals can increase anterior ground reaction forces (AGRF) unilaterally for the targeted limb. Thus, AGRF biofeedback may be a beneficial strategy to target unilateral propulsive deficits in people post-stroke. Incorporation of gaming interfaces for gait biofeedback can increase patient motivation, distract participants from fatigue or boredom, and encourage greater numbers of repetitions during gait training.

The long-term goal of this study is to develop a more engaging, motivating gait biofeedback methodologies specifically designed for post-stroke gait training. The researchers aim to address a major challenge for rehabilitation clinicians - to make gait training appealing and meaningful so that patients engage in sufficient repetitions, intensity, and challenge to maximize therapeutic effectiveness. The study premise is that post-stroke individuals will demonstrate greater engagement, motivation, and therapeutic benefits during gait training sessions involving biofeedback when training incorporates intuitive, entertaining, game-based interfaces. Outcomes of the study will include measures of participant engagement, user-reports and survey-responses on motivation, fatigue, game characteristics, and adverse effects (e.g. nausea, dizziness) during game exposure. In addition to this clinical trial with stroke survivor participants, data about the game interface will be collected by having able-bodied neuro-rehabilitation clinicians try the 2 types of biofeedback interventions.

Study participants will complete one sessions comprising exposure to gait biofeedback systems in a randomized order. Participants will be exposed to 2 types of biofeedback interfaces: (i) newly developed game-based interface (projector screen display), and (ii) traditional, non-game interface.

ELIGIBILITY:
Inclusion Criteria for Post-Stroke Participants:

* age 30 to 90 years
* chronic stroke (>6 months post stroke) affecting the right leg
* ambulatory with or without the use of a cane or walker
* able to walk for 2 minutes at the self-selected speed without an orthoses
* resting heart rate 40-100 beats per minute

Exclusion Criteria for Post-Stroke Participants:

* cerebellar signs (ataxic ("drunken") gait or decreased coordination during rapid alternating hand or foot movements)
* history of lower extremity joint replacement
* inability to communicate with investigators
* neglect/hemianopia, or unexplained dizziness in last 6 months
* neurologic conditions other than stroke
* orthopedic problems in the lower limbs or spine (or other medical conditions) that limit walking or cause pain during walking

Inclusion Criteria for Able-bodied Participants:

* age 18 to 90 years
* no history of neurologic disease
* no history of orthopedic disease or injury affecting the lower extremity

Exclusion Criteria for Able-bodied Participants:

* history of neurologic disease
* history of orthopedic disease or injury to the lower extremity in the past 6 months
* pain or discomfort during walking
* cardiovascular or medical condition affecting ability to exercise or walk

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Kesar, PT, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Rehabilitation Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results, after de-identification, will be available for sharing.
Time Frame: Individual participant data will be available for sharing beginning 9 months and ending 36 months after the article publication.
Access Criteria: Data will be available for sharing with investigators whose proposed used of the data has been approved by an independent review committee identified for this purpose. Data will be shared for the purposes of achieving the aims in the approved proposal. Proposals should be directed to trisha.m.kesar@emory.edu. To access the data, requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Alterman BL, Slusarenko A, Kim M, Alam Z, Fowler D, Krishnan S, Coleman MG, Wolf SL, Kesar TM. An innovative gamified gait biofeedback interface targeting propulsion: feasibility and preliminary effects. Res Sq [Preprint]. 2025 Dec 9:rs.3.rs-8099435. doi: 10.21203/rs.3.rs-8099435/v1. PMID 41510277

RESULTS

PARTICIPANT FLOW:
Groups:
- Post-stroke Participants: Post-stroke participants completing gait training trials with two different biofeedback interfaces in each experimental session. Participants also complete a control condition where no biofeedback is provided.
  AGRF Biofeedback Game: During the AGRF biofeedback game participants walk on a split-belt treadmill with a projector or screen display. Participants receive real-time information or feedback about ongoing gait performance parameters while they are walking. The participants are exposed to the AGRF biofeedback game for 4 minutes.
  Traditional Biofeedback Interface: For the traditional non-game biofeedback, the visual display comprises a horizontal line graph with a moveable cursor that represents the current measured value of antero-posterior ground reaction force for the targeted leg. The auditory feedback comprises an audible "beep" produced every time the cursor entered the target range. Participants are exposed to the traditional biofeedback interface for 4 minutes.
  Control Condition: Participants complete a control walk with out feedback.
- Able-bodied Participants: Able-bodied individuals completing gait training trials with two different biofeedback interfaces in each experimental session. Participants also complete a control condition where no biofeedback is provided.
  AGRF Biofeedback Game: During the AGRF biofeedback game participants walk on a split-belt treadmill with a projector or screen display. Participants receive real-time information or feedback about ongoing gait performance parameters while they are walking. The participants are exposed to the AGRF biofeedback game for 4 minutes.
  Traditional Biofeedback Interface: For the traditional non-game biofeedback, the visual display comprises a horizontal line graph with a moveable cursor that represents the current measured value of antero-posterior ground reaction force for the targeted leg. The auditory feedback comprises an audible "beep" produced every time the cursor entered the target range. Participants are exposed to the traditional biofeedback interface for 4 minutes.
  Control Condition: Participants complete a control walk with out feedback.
Period: Overall Study
Arm/Group | Post-stroke Participants | Able-bodied Participants
Started | 9 | 10
Completed | 7 | 9
Not Completed | 2 | 1
Not completed — Treadmill speed less than 0.50 miles per hour | 2 | 0
Not completed — Missing biomechanical data | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population includes participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Post-stroke Participants | Able-bodied Participants | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.43 (7.46) | 27.89 (4.14) | 43.44 (19.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Peak AGRF
Description: Paretic leg (right leg for post-stroke participants) or targeted leg (right leg for able-bodied participants) peak push off force (peak AGRF) was calculated from GRF data. Higher values indicate greater push off force.
Time Frame: After each biofeedback interface session on Day 1
Population: This analysis includes participants who completed the trial and had the right leg studied. One post-stroke participant had their left side affected and was not included in this analysis.
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Post-stroke Participants | Able-bodied Participants
Number analyzed (Participants) | 6 | 9
Newtons
  Traditional Biofeedback Interface | 99.1 (23.5) | 143.8 (62.1)
  AGRF Biofeedback Game | 95.6 (29.9) | 166.6 (67.4)

2. Primary Outcome: Trailing Limb Angle (TLA)
Description: The trailing limb angle contributes to increased propulsion during walking. Trailing limb angle is a kinematic variable derived from 3-dimensional motion capture, which measures the orientation of the leg with respect to the center of mass at the stance to swing transition. In stroke survivors, trailing limb angle increases as walking speed increases.
Time Frame: After each biofeedback interface session on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Post-stroke Participants | Able-bodied Participants
Number analyzed (Participants) | 6 | 9
degrees
  Traditional Biofeedback Interface | 19.56 (2.95) | 22.52 (3.06)
  AGRF Biofeedback Interface | 18.63 (2.69) | 24.22 (4.30)

3. Secondary Outcome: Likert Enjoyment/Boredom Scale Domain Scores
Description: The Likert Enjoyment Boredom Scale is a 4-item instrument evaluating user reports of perceived effort in four different domains: Enjoyment/Fun, Boredom, Motivation, and Challenge. To assess each domain, participants are asked:
  * How much enjoyment/fun did you feel in the previous walking trial?
  * How much boredom did you feel in the previous walking trial?
  * How much motivation did you feel in the previous walking trial?
  * How much challenge did you feel in the previous walking trial?
  Each question is scored on a 8-point scale from 1 to 8, where the intensity of each domain is scored as 1 = not at all to 8 = very much/a lot. For the individual domains, higher scores are interpreted as the participant experiencing greater enjoyment/fun, boredom, motivation, or challenge.
Time Frame: Day 1, after each of the biofeedback interface sessions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-stroke Participants | Able-bodied Participants
Number analyzed (Participants) | 7 | 9
score on a scale
  Enjoyment/Fun Domain Score for Traditional Biofeedback Interface | 5.57 (1.62) | 4.78 (2.33)
  Enjoyment/Fun Domain Score for AGRF Biofeedback Game | 6.29 (0.95) | 5.78 (0.97)
  Boredom Domain Score for Traditional Biofeedback Interface | 6.57 (2.30) | 5.22 (2.33)
  Boredom Domain Score for AGRF Biofeedback Game | 5.57 (2.37) | 6.56 (1.67)
  Motivation Domain Score for Traditional Biofeedback Interface | 6.86 (1.21) | 6.33 (1.41)
  Motivation Domain Score for AGRF Biofeedback Game | 6.71 (1.11) | 6.22 (1.79)
  Challenge Domain Score for Traditional Biofeedback Interface | 5.71 (1.50) | 4.11 (1.36)
  Challenge Domain Score for AGRF Biofeedback Game | 6.86 (1.07) | 6.00 (1.73)

4. Secondary Outcome: NASA Task Load Index (NASA - TLX)
Description: The NASA task load index (NASA - TLX) evaluates user reports of perceived effort in six subscales of Mental Demand, Physical Demand, Temporal Demand, Performance, Effort, and Frustration. Each subscale is scored on a 21-point scale from 1 to 21, where very low demand/perfect performance = 1 and very high demand/failure = 21. A total score is created by taking the average of each subscale; the total score ranges from 1 to 21 with higher scores indicating that the task is very demanding to perform.
Time Frame: Day 1, after each of the biofeedback interface sessions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-stroke Participants | Able-bodied Participants
Number analyzed (Participants) | 7 | 9
score on a scale
  Traditional Biofeedback Interface | 7.98 (1.87) | 6.89 (2.02)
  AGRF Biofeedback Game | 9.76 (2.75) | 10.83 (2.95)

5. Secondary Outcome: Borg Rating of Perceived Exertion (RPE) Scale
Description: The Borg Rating of Perceived Exertion (RPE) Scale asks respondents to report how hard it feels like their body is working with a single item. Perceived exertion is rated on a scale from 6 to 20 where "no exertion at all" is scored as 6 and "maximal exertion" is scored as 20. Ratings between 12 and 14 are generally considered as a moderate intensity level.
Time Frame: Day 1, during each of the biofeedback interface sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Post-stroke Participants | Able-bodied Participants
Number analyzed (Participants) | 7 | 9
units on a scale
  Traditional Biofeedback Interface | 10.29 (2.14) | 8.67 (1.22)
  AGRF Biofeedback Game | 10.43 (2.99) | 10.11 (3.33)

6. Secondary Outcome: User Evaluation Questionnaire (UEQ) Score
Description: User experience of the biofeedback game is assessed with a 26-item user evaluation questionnaire (UEQ). Participants indicate how they found the session to be for a variety of usability qualities, including likability, speed, and meeting expectations. Responses are given on a 7-point scale where scale where 1 = the most agreement with the adjective on the left, 4 = a neutral response, and 7 = the most agreement with the adjective on the right. For some items high scores are associated with positive perceptions, while for other items low low scores are associated with positive perceptions. Items were grouped according to whether high or low scores meant positive perceptions and separate summary scores were obtained by calculating the mean score for the items included, so that the summary scores range from t to 7.
Time Frame: Day 1, after each of the biofeedback sessions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-stroke Participants | Able-bodied Participants
Number analyzed (Participants) | 7 | 9
score on a scale
  Traditional Biofeedback Interface -Items Where High Score Value Indicates Positive Perceptions | 5.46 (0.75) | 5.19 (0.73)
  AGRF Biofeedback Game - Items Where High Score Value Indicates Positive Perceptions | 5.36 (1.20) | 5.41 (0.71)
  Traditional Biofeedback Interface -Items Where Low Score Value Indicates Positive Perceptions | 2.27 (0.55) | 2.69 (0.65)
  AGRF Biofeedback Game - Items Where Low Score Value Indicates Positive Perceptions | 2.36 (0.87) | 2.38 (0.66)

7. Other Pre Specified Outcome: Qualitative Feedback
Description: User experiences about the feedback will be obtained in the form of subjective comments.
Time Frame: Day 1, after each of the biofeedback sessions
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Heart Rate
Description: Participants wear a heart rate monitor placed on the chest under clothing (Polar USA, Lake Success ,NY) and heart rate is collected after every sixty seconds of walking.
Time Frame: Day 1, during and after each of the biofeedback sessions
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Skin Impedance
Description: A galvanic skin resistance (GSR) device is wrapped around the index and middle finger on the subject's left or right hand ensuring it was not on the bone of the fingers nor tightly wrapped to avoid blood flow restriction. These data are collected for 3 minutes when the subject is presented with the biofeedback interface.
Time Frame: Day 1, during each of the biofeedback sessions
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information about adverse events was collected during the biofeedback sessions on Day 1 of the study.
Arm/Group | Post-stroke Participants | Able-bodied Participants
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT04013971/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT04013971/ICF_000.pdf